CLINICAL TRIAL: NCT04750850
Title: The Effectiveness of Core Stability Exercises to Improve Balance and Gait in Hereditary Ataxias. Pilot Study
Brief Title: Core Stability Exercises and Hereditary Ataxia
Acronym: Core-ataxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Collaborators: Universitat de Lleida (Other)
Responsible Party: Principal Investigator, Rosa Cabanas Valdés, PhD, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Core protocol 1
Record Dates: First submitted 2021-02-10; First posted 2021-02-11 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Hereditary Ataxia; Spinocerebellar Degenerations; Cerebellar Ataxia
Keywords: ataxia; balance; gait ataxia; activities of daily living; core stability exercises; postural balance
MeSH Terms: conditions — Spinocerebellar Degenerations; Cerebellar Ataxia; Ataxia; Gait Ataxia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core stability exercises group (Experimental): 30 minutes of core stability exercises program at a light intensity and take a rest breaks if is necessary. They will be instructed in the use of the 4-5 points of the Borg 10 Rating of Perceived Exertion for self-monitoring of exercise intensity. The exercises will performed twice a day for 5 days a week during 5 weeks. A physiotherapist conducted an initial home visit to ensure correct execution of the exercises. He or she will teach the exercises and then the patient will perform them alone in your home. Once a week the physiotherapist will phone the patient and will ask her/him for doubts.
  Interventions: Other: Therapeutic core stability exercises
- Control group (Active Comparator): The patients to continue as normal and not change their routine in terms of exercise and physical activity during the period of study.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Therapeutic core stability exercises — exercises focused on trunk muscle strengthening, proprioception, selective movements of the trunk and pelvis muscle, and coordination, and will be carried out in supine, sitting on a stable surface and sitting on an unstable surface (ball). The exercise involves changes in the position of the body with or without resistance, aiming to improve strength, endurance, proprioception and coordination. Training is determined by the patient's ability to undertake easy exercises and progress to more challenging exercises.
  Other Names: trunk exercises
  Arms: Core stability exercises group
Other: Usual care — Usual routine as walking and activities of daily living.
  Other Names: Conventional physiotherapy
  Arms: Control group

SUMMARY:
The hereditary ataxias are a group of genetic disorders characterized by slowly progressive incoordination of gait and balance impairments in sitting and standing. Trunk local stability during gait is lower in patients with degenerative ataxia than that in healthy adult population.

Given the fact that drug interventions are rare in degenerative diseases and limited to only specific type of diseases and symptoms, physiotherapy is a major cornerstone in current therapy of ataxic gait. Core stability exercises training could be included as an adjunct to conventional balance training in improving dynamic balance and gait. Due to the nature of the interventions, the study will have a single blind design.

DETAILED DESCRIPTION:
The hereditary ataxias are a group of genetic disorders characterized by slowly progressive incoordination of gait and often associated with poor coordination of hands, speech, and eye movements. Prevalence of the autosomal dominant cerebellar ataxias (ADCAs) is estimated to be approximately 1-5:100,000 populations. Hereditary ataxia may result from: dysfunction of the cerebellum and its associated system, lesions in the spinal cord and/or peripheral sensory loss.

Clinical manifestations of hereditary ataxia are poor coordination of movement and a wide-based, uncoordinated, unsteady gait. Poor coordination of the limbs and of speech (dysarthria) are often present. Ataxia patients perceive impairments in balance, coordination and speech as the symptoms with greatest impact, as well as fatigue.

Postural disorders in cerebellar ataxia constitute a major cause of poor balance. Local stability of the trunk during gait in patients with cerebellar degenerative ataxia is lower than that in controls. To compensate for this instability, walkers increase the width of the base of support, take smaller steps and increase the duration of foot contact to the floor, sacrificing swing phase. They progress forward slower, with a lower cadence and preferred walking pace. This lack of stability is in turn correlated with the history of falls. Local stability of the trunk may thus be useful when planning gait and balance rehabilitation in patients with ataxia. Developing core strength is essential for everyday health and well-being, as a strong core protects the spine, reduces back pain, enhances movement patterns, and improves balance, stability and posture. However, while motor training programs have been shown to be beneficial in other neurodegenerative diseases (e.g., Parkinson's disease or stroke, their effectiveness remains controversial in the field of degenerative hereditary ataxias.

There's emerging evidence that rehabilitation may improve function, mobility, ataxia and balance in genetic degenerative ataxia. Although these conclusions are based primarily on moderate to low-quality studies, the consistency of positive effects verifies that rehabilitation is beneficial. Intensive rehabilitation (with balance and coordination exercises) improves the patients' functional abilities (level of proof: moderate). Although techniques such as virtual reality, biofeedback, treadmill exercises with supported body weight and torso weighting appear to be of value, their specific efficacy has yet to be characterized. This body of literature is limited by the wide range of underlying conditions studied and methodological weaknesses (small sample sizes, poorly described rehabilitation protocols, etc.

The aim of this study is that a program of core stability exercises could improve sitting and standing balance and gait in hereditary ataxia patients. Secondary objectives are activities of daily living, lower limb strength and health status of quality of life. After giving informed consent, participants will be randomly assigned (at a ratio 1:1) to core stability group or control group. Concealed treatment allocation will be performed via opaque envelopes.

The study will be carried out in accordance with the principles enunciated in the current version of the Declaration of Helsinki and the requirements of Spanish law and the Spanish regulatory authority.

ELIGIBILITY:
* Inclusion criteria: suffer a degenerative hereditary ataxia. spinocerebellar ataxia (SCA), Friedreich's ataxia (FRDA), idiopathic sporadic cerebellar ataxia, and specific neurodegenerative disorders in which ataxia is the dominant symptom (e.g. cerebellar variant of multiple systems atrophy (MSA-C). Both sexes and age ≥ 18 years old. •Ability to understand and execute simple instructions.
* Exclusion Criteria: Concurrent neurologic disorder (e. g. Parkinson's disease) or major orthopedic problem (e. g. amputation) that hamper sitting balance, relevant psychiatric disorders that may prevent from following instructions, Other treatments that could influence the effects of the interventions, Contraindication to physical activity (e.g., heart failure).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Rate of dynamic sitting balance and trunk coordination | T1: Baseline, T2: 5 weeks and T3: follow up 5 weeks
  Spanish-version of Trunk Impairment Scale 2.0. Each item will be performed three times and the highest score counts. Otherwise, no practice session allowed. The patient can be corrected between attempts. The tests are verbally explained to the patient and can be demonstrated if needed. There are two subscales: dynamic sitting balance and coordination. The first have 10 items and second 6. The highest possible total score is consequently 16 points, which indicates a good dynamic sitting balance and correct trunk control and sitting coordination. If the patient cannot maintain a sitting position for 10 seconds without back and arm support, with hands on thighs, feet in contact with the ground and knees bent at 90° (starting position), the total score for the scale is 0 points.
Rate of static sitting balance | T1: Baseline, T2: 5 weeks and T3: follow up 5 weeks
  Sitting section of Scale for the assessment and rating of ataxia (SARA). Patient is asked to sit on an examination bed without support of feet, eyes open and arms outstretched to the front. 0 Normal, no difficulties sitting >10 seconds, 1 Slight difficulties, intermittent sway, 2 Constant sway, but able to sit > 10 s without support, 3 Able to sit for > 10 s only with intermittent support, 4 Unable to sit for >10 s without continuous support
Rate of ataxia severity | T1: Baseline, T2: 5 weeks and T3: follow up 5 weeks
  Scale for the Assessment and Rating of Ataxia (SARA). The scale is made up of 8 items related to gait, stance, sitting, speech, finger-chase test, nose-finger test, fast alternating

SECONDARY OUTCOMES:
Rate of standing balance | T1: Baseline, T2: 5 weeks and T3: follow up 5 weeks
  Standing section of Scale for the assessment and rating of ataxia (SARA). Patient is asked to stand (1) in natural position, (2) with feet together in parallel (big toes touching each other) and (3) in tandem (both feet on one line, no space between heel and toe). Proband does not wear shoes, eyes are open. For each condition, three trials are allowed. Best trial is rated. 0 Normal, able to stand in tandem for > 10 seconds 1 Able to stand with feet together without sway, but not in tandem for > 10s, 2 Able to stand with feet together for > 10 s, but only with sway, 3 Able to stand for > 10 s without support in natural, position, but not with feet together, 4 Able to stand for >10 s in natural position only with intermittent support, 5 Able to stand >10 s in natural position only with constant support of one arm, 6 Unable to stand for >10 s even with constant support of one arm.
Rate of gait ability | T1: Baseline, T2: 5 weeks and T3: follow up 5 weeks
  Gait section of Scale for the assessment and rating of ataxia (SARA). Patient is asked (1) to walk at a safe distance parallel to a wall including a half-turn (turn around to face the opposite direction of gait) and (2) to walk in tandem (heels to toes) without support. Scoring items from 0 to 8: 0 Normal, no difficulties in walking, turning and walking tandem (up to one misstep allowed) and 8 Unable to walk, even supported.
  Gait speed by 4 meters walking test (meters per second) . The individual walks without assistance for 6 meters, with the time measured for the intermediate 4 meters to allow for acceleration and deceleration.
Rate of balance confidence | T1: Baseline, T2: 5 weeks and T3: follow up 5 weeks
  Activities-specific Balance Confidence (ABC). Larger typeset should be used for self-administration, while an enlarged version of the rating scale on an index card will facilitate in-person interviews. The ABC is an 11-point scale and ratings should consist of whole numbers (0-100) for each item. Total the ratings (possible range = 0 - 1600) and divide by 16 to get each subject's ABC score. If a subject qualifies his/her response to items #2, #9, #11, #14 or #15 (different ratings for "up" vs. "down" or "onto" vs. "off"), solicit separate ratings and use the lowest confidence of the two (as this will limit the entire activity, for instance the likelihood of using the stairs.) • 80% = high level of physical functioning
  • 50-80% = moderate level of physical functioning • < 50% = low level of physical, functioning . < 67% = older adults at risk for falling; predictive of future fall.
Rate of lower limb strength | T1: Baseline, T2: 5 weeks and T3: follow up 5 weeks
  30 seconds sit-to-stand. The 30-second chair stand involves recording the number of stands a person can complete in 30 seconds rather then the amount of time it takes to complete a pre-determined number of repetitions. That way, it is possible to assess a wide variety of ability levels with scores ranging from 0 for those who can not complete 1 stand to greater then 20 for more fit individuals.
Rate of adherence | T2: 5 weeks
  Adherence to the core stability exercise programme will be determined using exercise diaries, and process evaluation will be conducted via structured interviews with each participant at end of treatment.
Rate of health status | T1: Baseline, T2: 5 weeks and T3: follow up 5 weeks
  Health status by Euroqol 5 dimensions (EQ-5D). EQ-5D is a visual analogue scale for health ranging from 0 (worst possible) to 100 (best possible).
Rate of gait speed | T1: Baseline, T2: 5 weeks and T3: follow up 5 weeks
  4 meters walking test (4-MWT)
Rate of quality of life | T1: Baseline, T2: 5 weeks and T3: follow up 5 weeks
  Quality of life by EQ-5D-5L. The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression

CONTACTS AND LOCATIONS:
Overall Officials: Rosa C Cabanas-Valdés, PhD, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- Rosa Cabanas Valdés, Cardedeu, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen DH, Latimer C, Yagi M, Ndugga-Kabuye MK, Heigham E, Jayadev S, Meabon JS, Gomez CM, Keene CD, Cook DG, Raskind WH, Bird TD. Heterozygous STUB1 missense variants cause ataxia, cognitive decline, and STUB1 mislocalization. Neurol Genet. 2020 Feb 10;6(2):1-13. doi: 10.1212/NXG.0000000000000397. eCollection 2020 Apr. PMID 32211513
- [Background] Ruano L, Melo C, Silva MC, Coutinho P. The global epidemiology of hereditary ataxia and spastic paraplegia: a systematic review of prevalence studies. Neuroepidemiology. 2014;42(3):174-83. doi: 10.1159/000358801. Epub 2014 Mar 5. PMID 24603320
- [Background] OVERTON, Caroline E.; O'BRIEN, Kate. Guidelines on the Diagnosis and Management of Miscarriage. Early Pregnancy, 2017, 129.
- [Background] Marquer A, Barbieri G, Perennou D. The assessment and treatment of postural disorders in cerebellar ataxia: a systematic review. Ann Phys Rehabil Med. 2014 Mar;57(2):67-78. doi: 10.1016/j.rehab.2014.01.002. Epub 2014 Feb 6. PMID 24582474
- [Background] Chini G, Ranavolo A, Draicchio F, Casali C, Conte C, Martino G, Leonardi L, Padua L, Coppola G, Pierelli F, Serrao M. Local Stability of the Trunk in Patients with Degenerative Cerebellar Ataxia During Walking. Cerebellum. 2017 Feb;16(1):26-33. doi: 10.1007/s12311-016-0760-6. PMID 26811155
- [Background] Park J, Gong J, Yim J. Effects of a sitting boxing program on upper limb function, balance, gait, and quality of life in stroke patients. NeuroRehabilitation. 2017;40(1):77-86. doi: 10.3233/NRE-161392. PMID 27792020
- [Background] Cabanas-Valdes R, Urrutia G, Bagur-Calafat C, Caballero-Gomez FM, German-Romero A, Girabent-Farres M. Validation of the Spanish version of the Trunk Impairment Scale Version 2.0 (TIS 2.0) to assess dynamic sitting balance and coordination in post-stroke adult patients. Top Stroke Rehabil. 2016 Aug;23(4):225-32. doi: 10.1080/10749357.2016.1151662. Epub 2016 Mar 11. PMID 26922850
- [Background] Haruyama K, Kawakami M, Otsuka T. Effect of Core Stability Training on Trunk Function, Standing Balance, and Mobility in Stroke Patients. Neurorehabil Neural Repair. 2017 Mar;31(3):240-249. doi: 10.1177/1545968316675431. Epub 2016 Nov 9. PMID 27821673
- [Background] Cabrera-Martos I, Jimenez-Martin AT, Lopez-Lopez L, Rodriguez-Torres J, Ortiz-Rubio A, Valenza MC. Effects of a core stabilization training program on balance ability in persons with Parkinson's disease: a randomized controlled trial. Clin Rehabil. 2020 Jun;34(6):764-772. doi: 10.1177/0269215520918631. Epub 2020 Apr 29. PMID 32349543
- [Background] Cabanas-Valdes R, Bagur-Calafat C, Girabent-Farres M, Caballero-Gomez FM, Hernandez-Valino M, Urrutia Cuchi G. The effect of additional core stability exercises on improving dynamic sitting balance and trunk control for subacute stroke patients: a randomized controlled trial. Clin Rehabil. 2016 Oct;30(10):1024-1033. doi: 10.1177/0269215515609414. Epub 2015 Oct 8. PMID 26451007
- [Background] Synofzik M, Ilg W. Motor training in degenerative spinocerebellar disease: ataxia-specific improvements by intensive physiotherapy and exergames. Biomed Res Int. 2014;2014:583507. doi: 10.1155/2014/583507. Epub 2014 Apr 27. PMID 24877117
- [Background] He M, Zhang HN, Tang ZC, Gao SG. Balance and coordination training for patients with genetic degenerative ataxia: a systematic review. J Neurol. 2021 Oct;268(10):3690-3705. doi: 10.1007/s00415-020-09938-6. Epub 2020 Jun 24. PMID 32583055
- [Background] Milne SC, Corben LA, Georgiou-Karistianis N, Delatycki MB, Yiu EM. Rehabilitation for Individuals With Genetic Degenerative Ataxia: A Systematic Review. Neurorehabil Neural Repair. 2017 Jul;31(7):609-622. doi: 10.1177/1545968317712469. Epub 2017 Jun 9. PMID 28595509
- [Background] Seco, C. J., et al. Improvements in quality of life in individuals with friedreich's ataxia after participation in a 5-year program of physical activity: an observational study pre-post test design, and two years follow-up. Int J Neurorehabil, 2014, 1.3: 129
- [Background] Chang YJ, Chou CC, Huang WT, Lu CS, Wong AM, Hsu MJ. Cycling regimen induces spinal circuitry plasticity and improves leg muscle coordination in individuals with spinocerebellar ataxia. Arch Phys Med Rehabil. 2015 Jun;96(6):1006-13. doi: 10.1016/j.apmr.2015.01.021. Epub 2015 Feb 7. PMID 25668777
- [Background] Miyai I, Ito M, Hattori N, Mihara M, Hatakenaka M, Yagura H, Sobue G, Nishizawa M; Cerebellar Ataxia Rehabilitation Trialists Collaboration. Cerebellar ataxia rehabilitation trial in degenerative cerebellar diseases. Neurorehabil Neural Repair. 2012 Jun;26(5):515-22. doi: 10.1177/1545968311425918. Epub 2011 Dec 2. PMID 22140200
- [Background] Bunn LM, Marsden JF, Giunti P, Day BL. Training balance with opto-kinetic stimuli in the home: a randomized controlled feasibility study in people with pure cerebellar disease. Clin Rehabil. 2015 Feb;29(2):143-53. doi: 10.1177/0269215514539336. Epub 2014 Jul 31. PMID 25082955
- [Background] Velazquez-Perez L, Rodriguez-Diaz JC, Rodriguez-Labrada R, Medrano-Montero J, Aguilera Cruz AB, Reynaldo-Cejas L, Gongora-Marrero M, Estupinan-Rodriguez A, Vazquez-Mojena Y, Torres-Vega R. Neurorehabilitation Improves the Motor Features in Prodromal SCA2: A Randomized, Controlled Trial. Mov Disord. 2019 Jul;34(7):1060-1068. doi: 10.1002/mds.27676. Epub 2019 Apr 8. PMID 30958572
- [Background] Rodriguez-Diaz JC, Velazquez-Perez L, Rodriguez Labrada R, Aguilera Rodriguez R, Laffita Perez D, Canales Ochoa N, Medrano Montero J, Estupinan Rodriguez A, Osorio Borjas M, Gongora Marrero M, Reynaldo Cejas L, Gonzalez Zaldivar Y, Almaguer Gotay D. Neurorehabilitation therapy in spinocerebellar ataxia type 2: A 24-week, rater-blinded, randomized, controlled trial. Mov Disord. 2018 Sep;33(9):1481-1487. doi: 10.1002/mds.27437. Epub 2018 Aug 22. PMID 30132999
- [Background] Tabbassum, Khan Neha, et al. Core stability training with conventional balance training improves dynamic balance in progressive degenerative cerebellar ataxia. Indian Journal of Physiotherapy and Occupational Therapy, 2013, 7.1: 136.
- [Background] Schmitz-Hubsch T, du Montcel ST, Baliko L, Berciano J, Boesch S, Depondt C, Giunti P, Globas C, Infante J, Kang JS, Kremer B, Mariotti C, Melegh B, Pandolfo M, Rakowicz M, Ribai P, Rola R, Schols L, Szymanski S, van de Warrenburg BP, Durr A, Klockgether T, Fancellu R. Scale for the assessment and rating of ataxia: development of a new clinical scale. Neurology. 2006 Jun 13;66(11):1717-20. doi: 10.1212/01.wnl.0000219042.60538.92. PMID 16769946